CLINICAL TRIAL: NCT03328221
Title: A Pilot Observational Study of the Effects of Physical Activity on Heart Rate Variability in Patients With Severe Acquired Brain Injury
Brief Title: Physical Activity on Heart Rate Variability in Patients With Severe Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ingrid Poulsen, Director of research department RUBRIC, Rigshospitalet, Denmark
Other Study IDs: RH-2017-288, I-Suite: 05851
Record Dates: First submitted 2017-10-28; First posted 2017-11-01 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Acquired Brain Injury; Consciousness, Level Altered
Keywords: Heart rate variability; Observational study; Physical activity; Rehabilitation
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore autonomic cardiovascular regulation, through measures of heart rate variability (HRV), during different passive and active activities in patients with severe acquired brain injury and a low conscious state. Data from active rehabilitation will be compared with passive periods of rest as well as nightly variance during a continuous 5-day period.

DETAILED DESCRIPTION:
Background Severe acquired brain injury is usually associated with permanent disabilities in motor skills and cognitive functions that inhibit patients level of functioning, communication, participation in social activities and ability to work [Faul et al 2015, McLafferty et al 2016]. Patients with severe brain injury often have reduced level of consciousness in the early stages after the incident. Studies have shown that the autonomic nervous system can be affected in these patients, shown by analysis of the heart rate variability in the low frequency domain [Riberholt et al 2016, Vistisen et al 2014]. Signals from motor- and sensory cortex can influence sympathetic and parasympathetic activity and thus be a part of the cardiovascular adaptation during function [Sequeira et al 2000]. Aerobic exercise has been demonstrated to be effective regarding to autonomic cardiovascular regulation among healthy workers [Hallman et al 2017].

One method to assess sympathetic- and parasympathetic activity of the autonomous nervous system, as well as baroreflex sensitivity, is through the analysis of heart rate variability (HRV) [van de Vooren et al 2007]. A study of traumatic brain injured patients admitted to a neurocritical intensive care unit reveals that reduced HRV and baroreflex sensitivity within the first week of admission is associated with a poor neurological outcome at 1 year post-injury [Henden et al 2014]. Patients with severe acquired brain injury and low state of consciousness has demonstrated vastly reduced HRV and baroreflex sensitivity 40 days post injury during rest and head-up tilt[Riberholt et al 2016, Vistisen et al 2014].

Rehabilitation of patients with severe acquired brain injury and low state of consciousness is multimodal. Physical stimulation of the cardiovascular system can be exercised through an array of interventions such as mobilization, standing using a tilt-table, bed-biking, robot-assisted walking or other methods. To the authors' knowledge, no studies have been published researching the association between physical stimulation and HRV in patients with severe acquired brain injury in the subacute phase.

Hypotheses

* Patients with low state of consciousness have reduced HRV during rest.
* HRV is affected by physical activity such as, tilt-table mobilization, bed-biking or robot assisted walking.
* HRV is altered over time if patients are subjected to multiple bouts of physical exercise such as tilt-table mobilization, bed-biking or robot assisted walking.

Methods This is a prospective observational study. Patients are recruited from the Department of Neurorehabilitation/TBI Unit, Rigshospitalet, Denmark. This study will include patients above 18 years of age with severe acquired brain injury admitted for highly specialized neurorehabilitation. Patients must have a low level of consciousness defined as either vegetative or minimally conscious state. Five days of continuous heart rate monitorization at a sample rate of 256 Hz will start approximately 40 days after the initial injury using the ePatch® system. This study has been approved by the local ethics committee in the capital region of Denmark and oblige to the principles of the Helsinki Declaration. All data will be depersonalized and the Danish data protection agency has approved this study.

Treatment Participants will receive usual care, as practiced at the study location, regarding both medical care and rehabilitation efforts. There is no experimental intervention nor added or reduced treatment associated with this study.

Measurements Five days of continuous electrocardiography (ECG) will be recorded with ePatch (BioTelemetry Technology ApS, Denmark). The apparatus has a build-in inclinometer, accelerometer and the opportunity to mark the initiation of an event; in this case physical exercise, and is able to monitor heart rate continuously for five days at a sample rate of 256 Hz. The Epatch is attached to the patient's skin, over their sternum, using an adhesive patch. It can withstand most daily activities and is splash resistant. If medical imaging is necessary the ePatch will be removed and replaced afterwards.

Statistical analysis For statistical analysis of data comparing mean HRV of (T-exercise) with (T-rest) and (T-night) with (T-day) the paired t-test or equivalent non-parametric method will be utilized. A mixed effects model repeated measure analysis or equivalent non-parametric method (restricted maximum likelihood) will be performed for comparative analysis of variation from the 5 days of data collection.

Foreseeing the need in some cases to remove the ePatch, for various reasons, within the span of the 5 days of data collection, data will be included if events from 3 days of measurements can be extracted.

Data extracted from the participants medical record will be used to comprise a table of demographic characteristics that will include data on: age, sex, diagnose, body mass index (BMI), Glasgow Coma Score (GCS) at admittance, days removed from injury, level of functioning as measured with Early Functional Abilities scale (EFA) as well as level of consciousness as measured with Coma Recovery Scale - Revised (CRS-R). Likewise, data of participants medicinal intake during the study period will be retrieved from their medical record.

Ethical considerations As participants receive usual care no direct benefits are associated with this study.

Potential scientific benefits Researching autonomic cardiovascular regulation through HRV in patients with severe acquired brain injury is a relatively novel area. This exploratory study can help provide provisional information and thus generate further hypotheses for studies generating evidence of higher quality.

Harms The ePatch is designed for home-monitoring with an emphasis on ensuring minimum discomfort during use and is CE certified for clinical usage. During use or at removal, some individuals may experience slight skin-irritation under the adhesive patch that holds the ePatch in place. We assess the potential risks of participating in this study to be minimal.

Reporting of harms All adverse events related to participation in this study will be continuously monitored during the study. Besides notifying the local ethics committee, a list of encountered adverse events will be presented at publication.

Stopping guideline If 2 patients present allergic skin-reactions to the ePatch or adhesive patch during data collection the study will pause and consult with the manufacturers. If further 2 patients, after consultation with the manufacturers, present allergic skin-reactions the study will shut down.

Financial conditions This study is part of a thesis initiated by Jon Damsager Lauesen, Christian Gunge Riberholt and Karen Søgaard. Patients included in this study will not be financially compensated.

ELIGIBILITY:
Inclusion Criteria:

* Admitted at Department of Neurorehabilitation/TBI Unit, Rigshospitalet, Denmark
* Low conscious state (vegetative or minimally as determined by Glasgow Recovery Scale - Revised (CRS-R))

Exclusion Criteria:

* Known heart disease prior to brain injury
* Not possible to obtain informed consent
* Patients fiddling with or removing other monitoring equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted at Department of Neurorehabilitation/TBI Unit, Rigshospitalet, Denmark, with a low conscious state (vegetative or minimally conscious state) 40 days removed from injury.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Low frequency (LF) spectral analysis | 5 days of continuous measurements
  LF (0.05-0.15 Hz) during activity (T-exercise), rest (T-rest) and sleep (T-night)

SECONDARY OUTCOMES:
High frequency (HF) spectral analysis | 5 days of continuous measurements
  HF (0.15-0.35 Hz) during activity (T-exercise), rest (T-rest) and sleep (T-night)
LF/HF ratio | 5 days of continuous measurements
  The ratio between the power of LF and HF frequency bands during activity (T-exercise), rest (T-rest) and sleep (T-night)
SDRR | 5 days of continuous measurements
  Standard deviation of the RR-intervals during activity (T-exercise), rest (T-rest) and sleep (T-night)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Riberholt, Principal Investigator — Department of Neurorehabilitation, TBI Unit; Ingrid Poulsen, Study Director — Department of Neurorehabilitation, TBI Unit
Locations (1):
- at Department of Neurorehabilitation/TBI Unit, Rigshospitalet, Denmark, Copenhagen, Denmark

REFERENCES:
- [Background] Faul M, Coronado V. Epidemiology of traumatic brain injury. Handb Clin Neurol. 2015;127:3-13. doi: 10.1016/B978-0-444-52892-6.00001-5. PMID 25702206
- [Background] McLafferty FS, Barmparas G, Ortega A, Roberts P, Ko A, Harada M, Nuno M, Black KL, Ley EJ. Predictors of improved functional outcome following inpatient rehabilitation for patients with traumatic brain injury. NeuroRehabilitation. 2016 Jul 15;39(3):423-30. doi: 10.3233/NRE-161373. PMID 27589512
- [Background] Riberholt CG, Olesen ND, Thing M, Juhl CB, Mehlsen J, Petersen TH. Impaired Cerebral Autoregulation during Head Up Tilt in Patients with Severe Brain Injury. PLoS One. 2016 May 11;11(5):e0154831. doi: 10.1371/journal.pone.0154831. eCollection 2016. PMID 27168188
- [Background] Vistisen ST, Hansen TK, Jensen J, Nielsen JF, Fleischer J. Heart rate variability in neurorehabilitation patients with severe acquired brain injury. Brain Inj. 2014;28(2):196-202. doi: 10.3109/02699052.2013.860477. Epub 2013 Dec 2. PMID 24295072
- [Background] Sequeira H, Viltart O, Ba-M'Hamed S, Poulain P. Cortical control of somato-cardiovascular integration: neuroanatomical studies. Brain Res Bull. 2000 Sep 1;53(1):87-93. doi: 10.1016/s0361-9230(00)00312-9. PMID 11033212
- [Background] Hallman DM, Holtermann A, Sogaard K, Krustrup P, Kristiansen J, Korshoj M. Effect of an aerobic exercise intervention on cardiac autonomic regulation: A worksite RCT among cleaners. Physiol Behav. 2017 Feb 1;169:90-97. doi: 10.1016/j.physbeh.2016.11.031. Epub 2016 Nov 24. PMID 27889332
- [Background] van de Vooren H, Gademan MG, Swenne CA, TenVoorde BJ, Schalij MJ, Van der Wall EE. Baroreflex sensitivity, blood pressure buffering, and resonance: what are the links? Computer simulation of healthy subjects and heart failure patients. J Appl Physiol (1985). 2007 Apr;102(4):1348-56. doi: 10.1152/japplphysiol.00158.2006. Epub 2006 Dec 21. PMID 17185500
- [Background] Henden PL, Sondergaard S, Rydenhag B, Reinsfelt B, Ricksten SE, Aneman A. Can baroreflex sensitivity and heart rate variability predict late neurological outcome in patients with traumatic brain injury? J Neurosurg Anesthesiol. 2014 Jan;26(1):50-9. doi: 10.1097/ANA.0b013e3182a47b62. PMID 24064714